CLINICAL TRIAL: NCT06362395
Title: Ultra-high Dose Radiation for Liver Metastasis Using MR-guided TReatment With Stereotactic Ablative Single-fraction
Acronym: ULTRAS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-5022
Record Dates: First submitted 2024-02-26; First posted 2024-04-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Liver Metastases
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRL adaptive high dose (Experimental): Magnetic resonance (MR)-guided stereotactic ablative single-fraction with high dose radiation (27Gy)
  Interventions: Radiation: Magnetic resonance (MR)-guided stereotactic ablative single-fraction (SBRT)
- MRL adaptive ultra-high dose (Other): Magnetic resonance (MR)-guided stereotactic ablative single-fraction with ultra-high dose radiation (38Gy)
  Interventions: Radiation: Magnetic resonance (MR)-guided stereotactic ablative single-fraction (SBRT)

INTERVENTIONS:
Radiation: Magnetic resonance (MR)-guided stereotactic ablative single-fraction (SBRT) — Precise radiation therapy delivered in a single session using magnetic resonance imaging for guidance.

SUMMARY:
This international multi-centre phase 3 randomized control trial investigates whether giving a very high dose of radiation in a single treatment session (ultra-high dose: experimental) using advanced technology called MR-Linac is more effective than a high dose (control) for treating liver tumors that have spread from other parts of the body (liver metastases). This study also aims to identify predictors of treatment response and side effects by analyzing various factors such as imaging markers and genetic profiles.

Liver metastases are common in several cancers, but surgery is often not feasible for many patients. Stereotactic body radiotherapy (SBRT), which delivers focused radiation to tumors, is an alternative treatment option. Previous studies have shown promising results with SBRT, but the optimal radiation dose for liver metastases is still uncertain.

This study will look at patients with specific types of primary cancers known to respond well to SBRT. Treatment effectiveness will be assessed by monitoring tumor control, overall survival, and quality of life.

By comparing ultra-high dose SBRT with standard high dose, the study aims to determine if the former can provide better tumor control with fewer side effects. If successful, this approach could offer a significant advancement in the treatment of liver metastases, potentially improving outcomes and quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy (colorectal adenocarcinoma, pancreatic adenocarcinoma, head and neck SCC, cervix SCC, skin SCC and NSCLC) with metastatic liver disease detected on imaging. Biopsy of metastasis is preferred, but not mandatory.
* One, two or three liver metastases "target lesion", ≥ 2 cm from luminal and biliary structures
* Target lesions(s) that can receive high/ultra-high dose SBRT: Maximum number: 3, Maximum diameter of each target lesion: 6cm
* Non-target lesion(s) can be treated with single fraction SBRT with 16Gy or 24Gy, as soon as the total number of treated metastatic liver lesions with SBRT will be ≤5.
* Patients must be Child-Pugh score A within one month prior to study entry.
* Must be ≥ 18 years of age.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Expected life expectancy > 6 months.
* Suitable for MR-linac treatment (e.g., ability to lie on the treatment couch for at least one hour)
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in English. The baseline assessment must be completed within required timelines, prior to treatment start. Inability (lack of comprehension in English, or other equivalent reason such as cognitive issues or lack of competency) to complete the questionnaires will not make the patient ineligible for the study.
* Women of child bearing potential must use an accepted and effective method of contraception and/or abstain from sexual intercourse while on protocol treatment and for at least 6 months after the last day of RT. Sexually active males must use an accepted and effective method of contraception and/or abstain from sexual intercourse while on protocol treatment and for at least 6 months after SBRT.
* Women must not be pregnant or breast-feeding. All females of child bearing potential must have a serum or urine pregnancy test to rule out pregnancy within 4 weeks prior to registration. All breastfeeding women should discontinue breastfeeding prior to study registration.

Exclusion Criteria:

* Liver metastases from primary cancer other than listed in the eligibility criteria (i.e., tumor with low α/β ratio).
* Target lesion "planned for high/ultra-high dose SBRT" in proximity (<2cm) to luminal or biliary structures.
* Evidence of > 5 liver metastases (exception is in cases of oligoprogression, patients may have more than 5 liver metastases, but SBRT for target lesions will be required for 1, 2, or 3 liver metastases only).
* Any previous RT to the abdomino-pelvic region that would result in significant overlap of RT volume for the current study.
* Previous liver-directed transarterial radioembolization (note that previous transarterial chemoembolization, microwave ablation, or radiofrequency ablation are permitted).
* Individuals with severe, active co-morbidity including any of the following:
* Chronic obstructive pulmonary disease or other pulmonary illness requiring hospitalization within 30 days of study registration
* Unstable angina and/or congestive heart failure requiring hospitalization within the 30 days of study registration
* Acute myocardial infarction within 30 days of study registration
* Diseases precluding RT (e.g., active scleroderma, lupus or inflammatory bowel disease)
* Contraindications to MR imaging (e.g. implanted metallic prostheses, defibrillators, stimulators, pacemakers, or neurotransmitters) per institutional policy on management of patients with internal and external medical devices.
* History of claustrophobia
* The total length of treatment volume is beyond the capacity of MRL machine
* Participants must not be receiving any other standard anti-cancer therapy or experimental agent concurrently with SBRT (≥1 week break of systemic therapy prior to SBRT is required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Local control (LC) of treated target lesion compared to high dose MR-guided stereotactic single-fraction radiation. | 5 years
  The primary endpoint is LC defined as time from randomization to local failure of the treated target lesion. The LC will be estimated by cumulative incidence function with death and/or progression outside the treated target lesion (without local failure) as competing risk factors.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Endpoints related to patterns of failure, disease control, and survival will be determined by study investigators using standard-of-care imaging and clinical surveillance.
Progression free survival (PFS) | 5 years
  Endpoints related to patterns of failure, disease control, and survival will be determined by study investigators using standard-of-care imaging and clinical surveillance.
Intra-hepatic progression | 5 years
  Endpoints related to patterns of failure, disease control, and survival will be determined by study investigators using standard-of-care imaging and clinical surveillance.
Widespread progression. | 5 years
  Endpoints related to patterns of failure, disease control, and survival will be determined by study investigators using standard-of-care imaging and clinical surveillance.
Physician-assessed toxicities: National Cancer Institute (NCI) Common Terminology Criteria of Adverse Events (CTCAE) V.5. | 5 years
  Acute and late toxicities of treatment will be evaluated by CTCAE V5.0. The cumulative proportions of patients with at least one moderate to severe (grade 3-5) acute or late RT-related toxicity, measured by CTCAE (v5.0), will be compared between arms.
Patients-reported toxicity: Patient Reported Outcomes - Common Terminology Criteria of Adverse Events (PRO CTCAE) V.1. | 5 years
  Acute and late toxicities of treatment will be evaluated by PRO CTCAE (v1.0). The cumulative proportions of patients with at least one moderate to severe (grade 3-5) acute or late RT-related toxicity, measured by PRO CTCAE (v1.0), will be compared between arms.
Quality of life (QOL): European Organization for Research and Treatment of Cancer Quality of Life Questionnaires, Core 15 for Palliative Care (EORTC QLQ-C15-PAL) | Prior to treatment and after treatment up to 5 years.
  Acute and late toxicities of treatment will be evaluated by QOL (for English-speaking eligible patients) will be measured using the EORTC QLQ-C15-PAL, which will be administered before and after treatment. Scores of all domains of the EORTC questionnaires for each treatment arm will be evaluated before and after treatment.
Quality of life (QOL): European Organization for Research and Treatment of Cancer Quality of Life Questionnaires, liver metastases (EORTC QOQ-LM21). | Prior to treatment and after treatment up to 5 years.
  Acute and late toxicities of treatment will be evaluated by QOL (for English-speaking eligible patients) will be measured using the EORTC QOQ-LM21, which will be administered before and after treatment. Scores of all domains of the EORTC questionnaires for each treatment arm will be evaluated before and after treatment.

OTHER OUTCOMES:
Changes in the levels of circulating biomarkers (cell-free tumor DNA) in response to SBRT. | Before treatment, at 1 and 3 months post SBRT, and at disease progression
  Correlation analysis to determine the association between dynamic changes in biomarker levels and tumor response to SBRT and clinical outcomes. Biomarker analyses will be exploratory, involving various techniques such as quantitative analysis of circulating tumor DNA.
Changes in the levels of circulating biomarkers (cytokines) in response to SBRT. | Before treatment, at 1 and 3 months post SBRT, and at disease progression
  Correlation analysis to determine the association between dynamic changes in biomarker levels and tumor response to SBRT and clinical outcomes. Biomarker analyses will be exploratory, involving electrochemiluminescence assays for cytokine analysis.
Changes in the levels of circulating biomarkers (metabolites) in response to SBRT. | Before treatment, at 1 and 3 months post SBRT, and at disease progression
  Correlation analysis to determine the association between dynamic changes in biomarker levels and tumor response to SBRT and clinical outcomes. Biomarker analyses will be exploratory, involving liquid chromatography/mass spectrometry for metabolomics profiling.
Changes in the levels of circulating biomarkers (immune cell populations) in response to SBRT. | Before treatment, at 1 and 3 months post SBRT, and at disease progression
  Correlation analysis to determine the association between dynamic changes in biomarker levels and tumor response to SBRT and clinical outcomes. Biomarker analyses will be exploratory, involving flow cytometry analysis.
Identification of MR imaging biomarkers in response to SBRT. | 5 years
  Assessed through analysis of radiomic features from diagnostic and radiation therapy imaging datasets using MRI imaging analysis software.